CLINICAL TRIAL: NCT06703164
Title: Late Post Traumatic Ventriculomegally Does It Requires CSF Diversion ?
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nargis Samir Azmi Marqus, Resident Doctor, Assiut University
Other Study IDs: Post traumatic Hcp
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Hydrocephalus; Ventriculomegally
Keywords: Post Traumatic Hcp
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1 will be followed up by conservative management: This group will be followed up by close observation of GCS ,ct brain ,fundus examination &may need Csf flowmetry
- Group 2 will undergo csf diversion: Csf diversion is either vp shunt or evd

SUMMARY:
Aim of the study is :

1. prevelance of ventriculomegally in post traumatic patients after head trauma
2. To determine the incidence of surgically treated ventriculomegally within 6 months from head injury in a series of consecutive adult patients undergoing acute head CT following injury.
3. importance of csf diversion in post traumatic ventriculomegally

DETAILED DESCRIPTION:
Ventricular enlargement is a common finding after severe head injury.This is generally attributed to dysfunctional of perfusion and absorption of cerebrospinal fluid (CSF) or secondary to an atrophic process from neuronal loss.[ late post-traumatic ventriculomegally may be developed weeks to months after brain injury. Late post traumatic ventriculomegally incidence peaked within three months after injury .

Its incidence deeply varies among series (0.7-50%), and this is mainly due to very different diagnostic criteria Therefore, given the very high number of patients with traumatic brain injury (TBIs), patients presenting with late post-traumatic ventriculomegally are not infrequent.

The choice of the term ventriculomegally in the title reflects the difficulty in differentiating a ventricular enlargement (secondary to post-traumatic brain damage with atrophy) from an active hydrocephalic process.

Those patients with subarachnoid hemorrhage (SAH) had a threefold risk of developing ventriculomegally compared to patients with no SAH during the 2-year follow-up period. Also, decompressive craniectomy and the presence of subdural hygroma after craniectomy seem to increase the risk for ventriculomegally.In craniectomy, the proximity of the craniotomy to the skull midline might increase the risk as well. Other possible risk factors for post traumatic ventriculomegaly include: increased age, cerebrospinal fuid infection, and intraventricular hemorrhage . Inflammation-mediated adhesions related to intracranial hemorrhages can explain the predisposition to post traumatic ventriculomegally.

In fact, practically all patients with post-traumatic ventricular enlargement present with symptoms of post-taumatic Lesions and almost never present with the Hakim-adams trriad. Some of them present nonspecific symptoms, especially arrested clinical improvement during rehabilitation programs, impaired consciousness or a worsening neurologic status .

A classic clinical feature to suspect post traumatic ventriculomegally after TBI is poor improvement or stagnation of recovery .

Early recognition of post traumatic ventriculomegally is essential in the follow-up of patients with TBIs, as cerebrospinal fluid diversion (ventricular shunting) has been shown to improve outcome during rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* All post traumatic patients showing ventriculomegally in ct brain f/u (2week to 6months) after trauma.

Exclusion Criteria:

- 1.Any patient whose initial ct brain after head trauma showing ventriculomegally 2.any patient develops ventriculomegally within first 2 weeks of trauma or beyond 6 months of trauma.

3.any patient has hx of previous csf diversion .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ventricular enlargement is a common finding after severe head injury.[1] This is generally attributed to dysfunctional of perfusion and absorption of cerebrospinal fluid (CSF) or secondary to an atrophic process from neuronal loss.[2] late post-traumatic ventriculomegally may be developed weeks to months after brain injury. Late post traumatic ventriculomegally incidence peaked within three months after injury The choice of the term ventriculomegally in the title reflects the difficulty in differentiating a ventricular enlargement (secondary to post-traumatic brain damage with atrophy) from an active hydrocephalic process.
  A classic clinical feature to suspect post traumatic ventriculomegally after TBI is poor improvement or stagnation of recovery [11,12].
  Early recognition of post traumatic ventriculomegally is essential in the follow-up of patients with TBIs, as cerebrospinal fluid diversion (ventricular shunting) has been shown to improve outcome during rehabilitation [13,14].
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Late Post traumatic Ventriculomegally How frequently does it require csf diversion ? | From Dec 2024 to october 2025
  Ventricular enlargement is a common finding after severe head injury. This is generally attributed to dysfunctional of perfusion and absorption of cerebrospinal fluid (CSF) or secondary to an atrophic process from neuronal loss.
  late post-traumatic ventriculomegally may be developed weeks to months after brain injury. Late post traumatic ventriculomegally incidence peaked within three months after injury A classic clinical feature to suspect post traumatic ventriculomegally after TBI is poor improvement or stagnation of recovery .
  Early recognition of post traumatic ventriculomegally is essential in the follow-up of patients with TBIs, as cerebrospinal fluid diversion (ventricular shunting) has been shown to improve outcome during rehabilitation
Late Post traumatic Ventriculomegally How frequently does it require csf diversion ? | December 2024
  Ventricular enlargement is a common finding after severe head injury.This is generally attributed to dysfunctional of perfusion and absorption of cerebrospinal fluid (CSF) or secondary to an atrophic process from neuronal loss.
  late post-traumatic ventriculomegally may be developed weeks to months after brain injury. Late post traumatic ventriculomegally incidence peaked within three months after injury A classic clinical feature to suspect post traumatic ventriculomegally after TBI is poor improvement or stagnation of recovery.
  Early recognition of post traumatic ventriculomegally is essential in the follow-up of patients with TBIs, as cerebrospinal fluid diversion (ventricular shunting) has been shown to improve outcome during rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Elsayed mahmoud, Clinical Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De Bonis P, Mangiola A, Pompucci A, Formisano R, Mattogno P, Anile C. CSF dynamics analysis in patients with post-traumatic ventriculomegaly. Clin Neurol Neurosurg. 2013 Jan;115(1):49-53. doi: 10.1016/j.clineuro.2012.04.012. Epub 2012 May 15. PMID 22595485
- [Background] Shah AH, Komotar RJ. Pathophysiology of acute hydrocephalus after subarachnoid hemorrhage. World Neurosurg. 2013 Sep-Oct;80(3-4):304-6. doi: 10.1016/j.wneu.2013.01.110. Epub 2013 Feb 1. No abstract available. PMID 23376378
- [Background] Choi I, Park HK, Chang JC, Cho SJ, Choi SK, Byun BJ. Clinical factors for the development of posttraumatic hydrocephalus after decompressive craniectomy. J Korean Neurosurg Soc. 2008 May;43(5):227-31. doi: 10.3340/jkns.2008.43.5.227. Epub 2008 May 20. PMID 19096601
- [Background] Williams JR, Meyer MR, Ricard JA, Sen R, Young CC, Feroze AH, Greil ME, Barros G, Durfy S, Hanak B, Morton RP, Temkin NR, Barber JK, Mac Donald CL, Chesnut RM. Re-examining decompressive craniectomy medial margin distance from midline as a metric for calculating the risk of post-traumatic hydrocephalus. J Clin Neurosci. 2021 May;87:125-131. doi: 10.1016/j.jocn.2021.02.025. Epub 2021 Mar 20. PMID 33863519
- [Background] De Bonis P, Pompucci A, Mangiola A, Rigante L, Anile C. Post-traumatic hydrocephalus after decompressive craniectomy: an underestimated risk factor. J Neurotrauma. 2010 Nov;27(11):1965-70. doi: 10.1089/neu.2010.1425. PMID 20812777
- [Background] Lu VM, Carlstrom LP, Perry A, Graffeo CS, Domingo RA, Young CC, Meyer FB. Prognostic significance of subdural hygroma for post-traumatic hydrocephalus after decompressive craniectomy in the traumatic brain injury setting: a systematic review and meta-analysis. Neurosurg Rev. 2021 Feb;44(1):129-138. doi: 10.1007/s10143-019-01223-z. Epub 2019 Dec 16. PMID 31845199
- [Background] Fattahian R, Bagheri SR, Sadeghi M. Development of Posttraumatic Hydrocephalus Requiring Ventriculoperitoneal Shunt After Decompressive Craniectomy for Traumatic Brain Injury: a Systematic Review and Meta-analysis of Retrospective Studies. Med Arch. 2018 Jun;72(3):214-219. doi: 10.5455/medarh.2018.72.214-219. PMID 30061770
- [Background] Mazzini L, Campini R, Angelino E, Rognone F, Pastore I, Oliveri G. Posttraumatic hydrocephalus: a clinical, neuroradiologic, and neuropsychologic assessment of long-term outcome. Arch Phys Med Rehabil. 2003 Nov;84(11):1637-41. doi: 10.1053/s0003-9993(03)00314-9. PMID 14639563
- [Background] Hawkins TD, Lloyd AD, Fletcher GI, Hanka R. Ventricular size following head injury: a clinico-radiological study. Clin Radiol. 1976 Jul;27(3):279-89. doi: 10.1016/s0009-9260(76)80069-4. PMID 1086181
- [Background] Majdan M, Plancikova D, Brazinova A, Rusnak M, Nieboer D, Feigin V, Maas A. Epidemiology of traumatic brain injuries in Europe: a cross-sectional analysis. Lancet Public Health. 2016 Dec;1(2):e76-e83. doi: 10.1016/S2468-2667(16)30017-2. Epub 2016 Nov 29. PMID 29253420